CLINICAL TRIAL: NCT06521463
Title: WATCHMAN FLX™ Pro Left Atrial Appendage Closure Device With Alternative Post-Implant Monotherapy
Brief Title: SIMPLAAFY Clinical Trial
Acronym: SIMPLAAFY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S2508
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Stroke; Bleeding
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Aspirin (Experimental): Aspirin 81-100 mg, daily post implant for duration of the clinical trial
  Interventions: Device: WATCHMAN FLX Pro LAAC Device
- Reduced dose non-vitamin K antagonist (VKA) oral anticoagulant (NOAC) (Experimental): Reduced dose non-vitamin K antagonist (VKA) oral anticoagulant (NOAC) for the first 3 months daily, post implant, followed by aspirin only for the duration of the clinical trial
  Interventions: Device: WATCHMAN FLX Pro LAAC Device
- DAPT (Active Comparator): DAPT (aspirin 81-100 mg + clopidogrel 75 mg), for the first 6-months daily followed by aspirin only for the duration of the clinical trial
  Interventions: Device: WATCHMAN FLX Pro LAAC Device

INTERVENTIONS:
Device: WATCHMAN FLX Pro LAAC Device — WATCHMAN FLX Pro LAAC Device Implantation
  Other Names: WATCHMAN FLX Pro Left Atrial Appendage Closure Device

SUMMARY:
The primary objective is to demonstrate the safety and effectiveness of two monotherapy regimens versus dual antiplatelet (DAPT) therapy following post-implant with the WATCHMAN FLX Pro device in a commercial clinical setting.

DETAILED DESCRIPTION:
This study is a prospective, randomized, open-label, triple-arm, multi-center trial. Subjects will be randomized 1:1:1 to one of the three therapy arms and remain on treatment through the end of study (12 months):

1. Aspirin only
2. Reduced dose non-vitamin K antagonist (VKA) oral anticoagulant (NOAC)
3. DAPT

ELIGIBILITY:
Inclusion Criteria:

* Subject is of legal age to participate in the study per the laws of their respective geography.
* Subject is an acceptable candidate for a WATCHMAN FLX Pro device per the approved Instructions for Use.
* Subject is deemed to be suitable for all protocol defined drug regimens in the control and both test arms.
* The subject or legal representative is able to understand and willing to provide written informed consent to participate in the trial.
* The subject is able and willing to return for required follow-up visits and examinations.

Exclusion Criteria:

* Subject's device implant procedure was aborted (i.e., failed implant).
* Subject has a device margin residual leak > 0mm at time of implant.
* Occurrence of complications (major bleeding, systemic embolism, stroke, pericardial effusion requiring intervention) during the implant procedure, post-procedure, or prior to randomization.
* Subject has a contraindication to one of the three protocol defined drug regimens.
* Subject requires long-term anticoagulation therapy for reason other than AF-related stroke risk reduction or requires chronic P2Y12 inhibitor therapy.
* Subject has known history of severe liver disease including cirrhosis with a Child-Pugh classification C or D.
* Subject with known hypercoagulability disorder, mechanical heart valve, rheumatic heart disease, or recurrent deep vein thrombosis.
* Subject has intracardiac thrombus, LAA sludge, or dense spontaneous echo contrast (SEC) observed during pre-implant imaging.
* Subject has Modified Rankin Score of ≥ 3 at baseline.
* Subject has left ventricular ejection fraction (LVEF) < 30%.
* Subject with known amyloid cardiomyopathy.
* Platelet count ≤ 100,000 x 109/L.
* Subject has an estimated glomerular filtration rate (eGFR) < 30 ml/min (chronic kidney disease stage IV or V) or is on dialysis.
* Subject has a stroke (of any cause, whether ischemic or hemorrhagic) within 30 days prior to implant or prior to randomization.
* Subject has a documented myocardial infarction (MI) as either a non-ST elevation MI (NSTEMI) or as an ST-elevation MI (STEMI), with or without intervention, within 30 days prior to implant or prior to randomization.
* Subject had or is planning to have any cardiac or non-cardiac intervention or surgical procedure within 30 days prior to or 6-months after implant (including, but not limited to, cardioversion, percutaneous coronary intervention, cardiac ablation, cataract surgery, etc.).
* Subject has a major bleeding event per International Society on Thrombosis and Haemostasis (ISTH) definitions within the 30 days prior to implant or prior to randomization. Lack of resolution of related clinical sequelae or planned and pending interventions to resolve bleeding/bleeding source are a further exclusion regardless of timing of the bleeding event.
* Subject has an active bleed.
* Subject has a cardiac tumor.
* Subject has signs/symptoms of acute or chronic pericarditis.
* Subject has an active infection.
* There is evidence of tamponade physiology.
* Subject has New York Heart Association Class IV congestive heart failure at the time of implant or prior to randomization.
* Subject is currently enrolled in another investigational study, except if the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatment.
* Subject is of childbearing potential and is, or plans to become, pregnant during the time of the study.
* Subject has a documented life expectancy of less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1857 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Reduced dose NOAC Arm Primary Endpoint: Composite rate of all death, all stroke, systemic embolism, and ISTH major bleeding at 6-months after randomization in the reduced dose NOAC arm tested for non-inferiority compared to the DAPT arm | 6 months after randomization
  Non Inferiority
Aspirin Arm Primary Endpoint: Composite rate of all death, all stroke, systemic embolism, and ISTH major bleeding at 6-months after randomization in the Aspirin arm tested for non-inferiority compared to the DAPT arm. | 6 months after randomization
  Non Inferiority

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Saibal Kar, MD, Principal Investigator — Los Robles Health System; Walid Saliba, MD, Principal Investigator — The Cleveland Clinic
Locations (87):
- United States (87):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Grandview Medical Center, Birmingham, Alabama
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - HonorHealth Heart Group - Shea, Scottsdale, Arizona
  - Tucson Medical Center Healthcare, Tucson, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Mills Peninsula Health Services, Burlingame, California
  - John Muir Medical Center, Concord, California
  - Scripps Memorial Hospital, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - St. John's Health Center, Los Angeles, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - Cardiology Associates Medical Group, Ventura, California
  - Colorado Heart and Vascular PC, Lakewood, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Washington Hospital, Washington D.C., District of Columbia
  - Baptist Medical Center, Jacksonville, Florida
  - HCA Florida Mercy Hospital, Miami, Florida
  - Naples Community Hospital, Naples, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Georgia Arrhythmia Consultants, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Straub Medical Center, Honolulu, Hawaii
  - St. Luke's Boise Medical Center, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Evanston Hospital, Evanston, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Community Heart and Vascular Hospita, Indianapolis, Indiana
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Charlton Memorial, Fall River, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - M Health Fairview St John's Hospital, Maplewood, Minnesota
  - Mayo Clinic Foundation, Rochester, Minnesota
  - Centracare Heart and Vascular Center, Saint Cloud, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - St. Luke's Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital - University Medical Center, Camden, New Jersey
  - Virtua Health, Marlton, New Jersey
  - Valley Hospital, Paramus, New Jersey
  - Lovelace Medical Center, Albuquerque, New Mexico
  - Northwell Health, Bay Shore, New York
  - Kaleida Health, Buffalo, New York
  - New York University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Bethesda North Hospital-Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Legacy Emanuel Hospital & Health Center, Portland, Oregon
  - Pinnacle Health at Harrisburg Hospital, Harrisburg, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - Prisma Health, Columbia, South Carolina
  - MUSC Health Columbia Medical Center Downtown, Columbia, South Carolina
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - St. Thomas Heart, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - Orion Medical, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - Christus Trinity Mother Frances Health System-Hospital, Tyler, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Chippenham & Johnston-Willis Hospital, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Monongalia General Hospital, Morgantown, West Virginia
  - Bellin Health, Green Bay, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
URL: https://www.bostonscientific.com/content/gwc/en-US/data-sharing-requests.html